CLINICAL TRIAL: NCT06400173
Title: Validation Of The Flemish Montreal Cognitive Assessment (MoCA) For Persons With Hearing Impairment
Acronym: MoCA-HI
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: ONZ-2023-0147
Record Dates: First submitted 2024-04-12; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Dementia; Hearing Loss
Keywords: Cognitive screening; Montreal Cognitive Assessment
MeSH Terms: conditions — Dementia; Hearing Loss | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Individuals (>45 years) with mild cognitive impairment and hearing loss: All tests will be administered.
  Interventions: Behavioral: Cognitive screening; Behavioral: Audiological Assessment
- Individuals (>45 years) with dementia (Alzheimer, vascular or mixed) and hearing loss: All tests will be administered.
  Interventions: Behavioral: Cognitive screening; Behavioral: Audiological Assessment
- Individuals (>45 years) with age-normal cognition and hearing loss: All tests will be administered.
  Interventions: Behavioral: Cognitive screening; Behavioral: Audiological Assessment

INTERVENTIONS:
Behavioral: Cognitive screening — The Dutch Montreal Cognitive Assessment for persons with hearing loss (MoCA-HI) is a modified version of the original MoCA test specifically designed for individuals with hearing loss. It includes adaptations such as visual aids to accommodate for hearing loss, ensuring fair assessment of cognitive abilities in this population.
Behavioral: Audiological Assessment — Four audiological tests are included in the audiological assessment
  1. Tympanometry to assss the middle ear status
  2. Pure-tone audiometry with headphone to evaluate the hearing thresholds
  3. Speech audiometry in free field to assess the ability to understand spoken words in the presence of background noise
  4. The hAVICOP questionnaire to assess the hearing-related quality of life

SUMMARY:
The Montreal Cognitive Assessment (MoCA) is a screening test for detecting cognitive impairment that assesses several cognitive domains (attention and concentration, arithmetic and orientation, memory, etc.). The instructions as well as some test items of the MoCA are presented auditory (spoken). Consequently, performance on the MoCA may be co-dependent on hearing. Therefore, to rule out the possible negative influence of hearing loss on performance on the MoCA, a MoCA for individuals with hearing loss was recently developed. More specifically, the original MoCA was modified by providing the instructions audiovisually (spoken with visual support) as well as by replacing hearing-dependent items. Since replacing items may affect sensitivity and specificity, the MoCA for persons with hearing loss should be revalidated.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 60 years or older
* Individuals with normal vision (with lenses or glasses if needed)
* Individuals with age-related hearing loss
* Dutch-speaking individuals
* Individuals capable of giving consent to participate in the study themselves
* Individuals still residing in their own homes
* Individuals with an official diagnosis of dementia (Alzheimer's, vascular, or mixed) or mild cognitive impairment. This inclusion criterion applies only to the group with cognitive impairment.

Exclusion Criteria:

For individuals without cognitive impairment, the following exclusion criteria apply:

* (History of) neurological problems (brain tumor, epilepsy, history of stroke, etc.)
* Use of influencing medication (e.g., Ritalin and antidepressants)

Ages: 45 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals with cognitive impairment and/or hearing loss
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hearing status | This parameter will be assessed once during the first study visit of the patient. Test duration is approximately 20 minutes.
  Based on the results of the tympanometry and pure-tone audiometry the hearing status of the participant will be classified as normal or abnormal. In case of abnormal hearing, the type and severity will be specified.
MoCA-HI | This parameter will be assessed once (during the first study visit) or twice (during the second study visit 4 weeks later), depending on the random selection for the test-retest group. Test duration is approximately 15 minutes.
  The result (max 30) on the MoCA-HI will be calculated.
Hearing-related quality of life | This parameter will be assessed once during the first study visit of the patient. Test duration is approximately 15 minutes.
  Mean scores will be calculated for each subdomain separately (auditory-visual, cognitive, and psychosocial functioning) as well as combined within a total score. The scores can range from 0 to 100 whereby the worse one's hearing-related quality of life, the lower the score.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Van Langenhove, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Ghent Hospital, Ghent, East-Flanders, Belgium